CLINICAL TRIAL: NCT05776160
Title: Expanded Access Study for the Treatment of Patients With Commercially Out-of-Specification Axicabtagene Ciloleucel
Status: Available | Type: Expanded Access
Sponsor: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Other Study IDs: KT-US-471-0140; jRCT2033230370 (Other: Japan Registry of Clinical Trials)
Record Dates: First submitted 2023-03-03; First posted 2023-03-20 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Large B-cell Lymphoma; Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — axicabtagene ciloleucel

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Axicabtagene Ciloleucel — A single infusion of chimeric antigen receptor (CAR)-transduced autologous T cells/kg administered intravenously.
  Other Names: Yescarta®

SUMMARY:
The goal of this study is to provide access to axicabtagene ciloleucel for patients diagnosed with a disease approved for treatment with axicabtagene ciloleucel, that is otherwise out of specification for commercial release.

ELIGIBILITY:
Inclusion Criteria:

* Have commercially manufactured axicabtagene ciloleucel that does not meet commercial release criteria but does meet Kite clinical trial release criteria
* Females of childbearing potential must have a negative serum or urine pregnancy test (females who have undergone surgical sterilization or who have been post-menopausal for at least 2 years are not considered to be of childbearing potential)
* Deemed medically fit and stable to receive the product per the investigator's evaluation
* Repeat leukapheresis is not feasible per the investigator's assessment
* Be diagnosed with 1 of the approved labeled indications for axicabtagene ciloleucel that is intended for release
* In the investigator's opinion, there is no satisfactory alternative therapy available to the individual

Exclusion Criteria:

* History of severe immediate hypersensitivity to any drugs or metabolites of similar chemical classes as axicabtagene ciloleucel
* Uncontrolled active infection or inflammation per physician assessment
* Primary central nervous system lymphoma

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (121):
- United States (48):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - City of Hope Medical Center, Duarte, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Mayo Clinic Florida, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - St. Luke's Cancer Institute, Boise, Idaho
  - Northwestern Memorial Hospital, Chicago, Illinois
  - The University of Kansas Medical Center, Westwood, Kansas
  - University of Maryland Cancer Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute - Chestnut Hill, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine- Siteman Cancer Center, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Cornell Medicine - NewYork-Presbyterian Hospital, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center (MMC), The Bronx, New York
  - UNC Hospitals, The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center- James Cancer Hospital, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Vanderbilt-Ingrim Cancer Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Methodist Healthcare System of San Antonio dba Methodist Hospital, San Antonio, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - University of Virginia Comprehensive Cancer Center, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Japan (73):
  - Anjo Kosei Hospital, Aichi
  - Nagoya Medical Center, Aichi
  - Nagoya City University Hospital, Aichi
  - Aichi Medical University Hospital, Aichi
  - Akita University Hospital, Akita
  - Chiba University Hospital, Chiba
  - Ehime University Hospital, Ehime
  - University of Fukui Hospital, Fukui
  - Kokura Kinen Hospital, Fukuoka
  - Hamanomachi Hospital, Fukuoka
  - Kyushu Medical Center, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - Kurume University Hospital, Fukuoka
  - Gifu Municipal Hospital, Gifu
  - Gunma University Hospital, Gunma
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital, Hiroshima
  - Hiroshima University Hospital, Hiroshima
  - Sapporo Hokuyu Hospital, Hokkaido
  - Hokkaido University Hospital, Hokkaido
  - Kobe University Hospital, Hyōgo
  - Kobe City Medical Center General Hospital, Hyōgo
  - Hyogo Medical University Hospital, Hyōgo
  - University of Tsukuba Hospital, Ibaraki
  - Kagawa University Hospital, Kagawa
  - Kagoshima University Hospital, Kagoshima
  - Yokohama City University Medical Center, Kanagawa
  - Yokohama City University Hospital, Kanagawa
  - Kanazawa University Hospital, Kanazawa
  - Kumamoto University Hospital, Kumamoto
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Japanese Red Cross Kyoto Daiichi Hospital, Kyoto
  - Kyoto University Hospital, Kyoto
  - Mie University Hospital, Mie
  - Tohoku University Hospital, Miyagi
  - University of Miyazaki Hospital, Miyazaki
  - Shinshu University Hospital, Nagano
  - Nagasaki University Hospital, Nagasaki
  - Japanese Red Cross Aichi Medical Center Nagoya Daiichi Hospital, Nagoya
  - Nagoya University Hospital, Nagoya
  - Niigata University Medical & Dental Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Kurashiki Central Hospital, Okayama
  - Univercity of the Ryukyus Hospital, Okinawa
  - Osaka International Cancer Institute, Osaka
  - Osaka Red Cross Hospital, Osaka
  - Osaka Metropolitan University Hospital, Osaka
  - The University of Osaka Hospital, Osaka
  - Kansai Medical University Hospital, Osaka
  - Kindai University Hospital, Osaka
  - Oita University Hospital, Ōita
  - Jichi Medical University Saitama Medical Center, Saitama
  - Saitama Medical Center, Saitama
  - Shiga University of Medical Science Hospital, Shiga
  - Shimane University Hospital, Shimane
  - Hamamatsu University Hospital, Shizuoka
  - Jichi Medical University Hospital, Tochigi
  - Tokushima University Hospital, Tokushima
  - National Cancer Center Hospital, Tokyo
  - Toranomon Hospital, Tokyo
  - Jikei University Hospital, Tokyo
  - Juntendo University School of Medicine Juntendo Clinic, Tokyo
  - Institute of Science Tokyo Hospital, Tokyo
  - The University of Tokyo Hospital, Tokyo
  - Tokyo Metropolitan Cancer and Infectious diseases Center Komagome Hospital, Tokyo
  - Keio University Hospital, Tokyo
  - Teikyo University Hospital, Tokyo
  - Nihon University Itabashi Hospital, Tokyo
  - Tokyo Metropolitan Tama Medical Center, Tokyo
  - Tottori Univeristy Hospital, Tottori
  - Toyama Prefectural Central Hospital, Toyama
  - Wakayama Medical University Hospital, Wakayama
  - Yamagata University Hospital, Yamagata
  - Yamaguchi University Hospital, Yamaguchi

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT05776160